CLINICAL TRIAL: NCT04264455
Title: Evaluation of Long-term Incidence of Ventricular Arrhythmias in Patients With Acute Myocarditis
Acronym: AIM-ICD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: MVZ Leopoldina GmbH (Other); Brandenburg Medical School Theodor Fontane (Other); Hannover Medical School (Other)
Responsible Party: Principal Investigator, PD Dr. Peter Nordbeck, PD Dr. med. Peter Nordbeck, Wuerzburg University Hospital
Other Study IDs: IT-II-2019
Record Dates: First submitted 2019-12-19; First posted 2020-02-11 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Myocarditis Acute; Ventricular Arrythmia
Keywords: ICD; Life Vest; BioMonitor; Myocarditis; Ventricular Arrythmia
MeSH Terms: conditions — Myocarditis | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — hsTroponin T, CK, CK-MB, NT-proBNP, renal retention parameters, LDH, GOT, CRP, blood count, electrolytes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Biomonitor only: Patients receive a Biomonitor only
  Interventions: Device: Biomonitor; Device: Implantable Cardioverter-Defibrillator (ICD)
- Wearable Cardioverter-Defibrillator (Life Vest) + Biomonitor: Patients receive a Wearable Cardioverter-Defibrillator (Life Vest) combined with a Biomonitor
  Interventions: Device: Biomonitor; Device: Life Vest; Device: Implantable Cardioverter-Defibrillator (ICD)
- ICD Implantation: Patients receive an ICD only
  Interventions: Device: Implantable Cardioverter-Defibrillator (ICD)

INTERVENTIONS:
Device: Biomonitor — Patients receive a Biomonitor only
  Groups: Biomonitor only; Wearable Cardioverter-Defibrillator (Life Vest) + Biomonitor
Device: Life Vest — Patients receive a Wearable Cardioverter-Defibrillator; a Biomonitor is implanted additionally
  Groups: Wearable Cardioverter-Defibrillator (Life Vest) + Biomonitor
Device: Implantable Cardioverter-Defibrillator (ICD) — Patients receive an Implantable Cardioverter-Defibrillator (ICD)

SUMMARY:
Myocarditis is an inflammatory disease of the heart muscle which is mostly caused by viruses, bacteria, parasites, toxic substances/drugs or by primary autoimmune mechanisms. Signs of heart failure (dyspnea, reduced resilience, tendency to edema), thoracic pain, palpitations / arrhythmias / syncope, as well as (potentially) lethal clinical conditions in the sense of a cardiogenic shock or sudden cardiac death can be found.

In 2015, the European Society of Cardiology (ESC) gave a IIa recommendation for the indication of an ICD vest restoration as "bridging" until the acute phase subsides (possibly normalisation of the left ventricular pump function with reduced probability of malignant cardiac arrhythmia) or until ICD implantation in cases of severe LV dysfunction and/or ventricular electrical instability. The Monitoring and analysis of malignant cardiac arrhythmias are therefore crucial in the treatment of acute myocarditis.

The aim of this study is to observe the long-term incidence of ventricular arrhythmias in patients diagnosed with myocarditis and to analyze the MRI and echocardiographic data obtained as potential predictive factors for the occurrence of ventricular arrhythmias.

DETAILED DESCRIPTION:
Myocarditis is an inflammatory disease of the heart muscle, which is mostly caused by viruses, bacteria, parasites, toxic substances/drugs or by primary autoimmune mechanisms. In the first phase of acute myocarditis direct cell damage, in a second phase myocardial inflammation with additional myocardial damage can be observed. Symptoms vary widely and may include signs of heart failure (dyspnoea, reduced exercise capacity, edema tendency), chest pain, palpitations / arrhythmias / syncope, and (potentially) lethal clinical conditions such as cardiogenic shock or sudden cardiac death. Predictors of increased mortality are syncopes, malignant arrhythmias EF≤35% or heart failure NYHA III-IV. ICD implantation is recommended <3 months after manifestation only in exceptional situations (e.g. following resuscitation). The European Society of Cardiology (ESC) issued a IIa recommendation in 2015 for the indication of ICD vest fitting as "bridging" until the acute phase subsides (possible normalization of left ventricular pumping function with reduced probability of malignant cardiac arrhythmias) or until ICD implantation in cases of severe LV dysfunction and/or ventricular electrical instability is necessary. The observation, monitoring and analysis of malignant cardiac arrhythmias are therefore crucial in the treatment of acute myocarditis.

The aim of this study is to observe the long-term incidence of ventricular arrhythmias in patients with diagnosed myocarditis and to analyze the MRI and echocardiographic data obtained as potential predictive factors for the occurrence of ventricular arrhythmias.

The study is a prospective multicenter registry study. All potentially stressful measures and examinations such as blood sampling and echocardiography - except for follow-up MRI examinations - are carried out at our centre as standard clinical progress assessment, even independently of participation in the registry. The indication for biomonitor implantation is given after initial screening by means of a 24h-LZ-ECG with positive results (detection of ventricular arrhythmias). The registry study is performed with approved IECDs (Implantable electronic cardiovascular devices: Biomonitor (BioMonitor 2-AF, BioMonitor 3-AF (after release)), Biotronik® ICD) as well as WCD (Wearable Cardioverter Defibrillator, Zoll® LifeVest) and Biotronik® Cardio Messenger. The implantation is carried out exclusively according to the indication/testing guidelines. Thus, there are no risks or disadvantages for the participating patient.

The primary aim of the study is to monitor the long-term incidence of ventricular arrhythmias in patients with diagnosed myocarditis and to identify potential predictive factors for their occurrence.

Secondary goal is to analyze the long-term survival and need for heart transplantation and to identify MRI/echocardiographic parameters as determinants of arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* secured myocarditis via MRT / endomyocardial biopsy
* ventricular arrhythmias (≥ 5 beats) in the ECG / LZ ECG with clinical indication for a WCD system/ biomonitor/ or the indication for primary/secondary prophylactic ICD implantation
* presence of informed consent
* age >18 and <85 years

Exclusion Criteria:

* Participation in another study with an active treatment group
* Pregnant or breastfeeding women

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The groups will be selected from all patients attending the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Monitoring the change of long-term incidence of ventricular arrhythmias in patients with acute myocarditis at several follow-up dates. | 24 months follow-up
  The primary aim of the study is to monitor the long-term incidence of ventricular arrhythmias and/or sudden cardiac death in patients with diagnosed myocarditis and identify potential predictive factors for their occurrence.
  The 2-years incidence of sudden cardiac death and ventricular arrhythmias acquired by the respective device holters in use is investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nordbeck, MD, PhD, Principal Investigator — University Hospital Wuerzburg; Jonas Muentze, MD, Principal Investigator — University Hospital Wuerzburg
Locations (1):
- Wuerzburg University Hospital, Würzburg, Bavaria, Germany